CLINICAL TRIAL: NCT07296822
Title: A Randomized Controlled Trial of Internet-Based Cognitive Behavioral Therapy for MRI-Related Anxiety
Brief Title: Internet-Based Cognitive Behavioral Therapy for MRI-Related Anxiety
Acronym: MRTightxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johan Kihlberg (Other Government)
Collaborators: Linkoeping University (Other Government); Region Östergötland (Other); Region Jönköping County (Other Government); Landstinget i Kalmar Län (Other)
Responsible Party: Sponsor-Investigator, Johan Kihlberg, Associate Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EPM Dnr 2024-00435-01; Dnr 2024-00435-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2025-05-01; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Claustrophobia; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Anxiety Disorders; Claustrophobia | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The patients will undergo a four-week treatment that includes information about MRI, anxiety management, relaxation and retention. The end goal is to simulate an MRI scan in a mock scanner where participants can report their anxiety. Half of the participants will be randomized to receive the treatment before (intervention group) the simulated MRI scan and half will receive the treatment after the simulated MRI scan (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (No Intervention): Participants will receive the same iCBT intervention after completing the mock MR examination.
- Intervention (Experimental): Participants will receive the internet-based cognitive behavioral therapy (iCBT) intervention prior to undergoing the mock MR examination.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Participants will receive the internet-based cognitive behavioral therapy (iCBT) intervention prior to undergoing the mock MR examination.
  Arms: Intervention

SUMMARY:
The aim of the study is to investigate whether internet-based cognitive behavioural therapy (iCBT) can help patients who have difficulty undergoing magnetic resonance imaging (MRI). The main question to be answered is

- Can patients undergo MRI with less anxiety using iCBT?

The patients will undergo a four-week treatment that includes information about MRI, anxiety management, relaxation and retention. The end goal is to simulate an MRI scan in a mock scanner where participants can report their anxiety. Half of the participants will be randomized to receive the treatment before (intervention group) the simulated MRI scan and half will receive the treatment after the simulated MRI scan (control group). Up to 60 patients will be included plus some pilot patients.

ELIGIBILITY:
Inclusion Criteria:

* self-perceived problems with doing MRI examinations

Exclusion Criteria:

* difficulty understanding written text
* severe mental health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI-related anxiety | Baseline and within two days of the mock MRI examination
  MRI-related anxiety using the Magnetic Resonance Imaging Anxiety Questionnaire (MRI-AQ) measured before and after the mock MRI examination. Higher value means increased symptoms. Can give between 15-60 points.

SECONDARY OUTCOMES:
Anxiety | Baseline and within two days of the mock MRI examination
  Anxiety using Generalized Anxiety Disorder Seven Item Scale (GAD-7) measured before and after the mock MRI examination. Higher value means increased symptoms. Can give between 0-27 points.
Claustrophobia | Baseline and within two days of the mock MRI examination
  Claustrophobia using a Swedish validated translation of The Claustrophobia Questionnaire (CLQ) measured before and after the mock MRI examination. Higher value means increased symptoms. Can give between 0-48 points.
Mental health | Baseline and within two days of the mock MRI examination
  Mental health using the Patient Health Questionnaire-9 (PHQ-9) measured before and after the mock MRI examination. Higher value means increased symptoms. Can give between 0-27 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be stored at Linköping University, which the entire research group has full access to. No unauthorized persons will have access to the data.
  This is a research project with a quantitative method where the results are reported in aggregated form.
  The data is reported completely anonymized and only at the group level.

REFERENCES:
- See also: Study information for patients — https://www.iterapi.se/sites/tmri/
- See also: Study information — https://liu.se/forskning/mr-trangest